CLINICAL TRIAL: NCT04418713
Title: Active Video Games Against Obesity and Sedentarism in Children Between 9 and 11 Years Old: a Disruptive Proposal
Brief Title: Active Videogames Against Obesity in Children
Acronym: VIDEOACTIVO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad de Zaragoza (Other)
Responsible Party: Principal Investigator, José A. Casajús, Professor, Universidad de Zaragoza
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: DEP2017-85194-P
Record Dates: First submitted 2019-03-13; First posted 2020-06-05 (Actual); Last update posted 2024-01-12 (Actual); Status verified 2024-01

CONDITIONS: Childhood Obesity; Physical Activity; Sedentary Lifestyle; Body Fat
Keywords: Obesity; Sedentary Lifestyle; Physical Activity; Childhood Obesity; Exergames; Body Composition; Physical Fitness; Cardiometabolic Risk
MeSH Terms: conditions — Pediatric Obesity; Motor Activity; Sedentary Behavior; Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- exercise group with active video-games (Experimental): exergaming exercise: A combination of traditional exercise and exercise through active video games performed 3 days a week for one hour during 7 months. As well, it will be including some session about nutritional advice.
  Interventions: Other: active video-games
- control group (No Intervention): no physical intevention will be provided, but it will be included some sessions on nutritional advice.

INTERVENTIONS:
Other: active video-games — An intervention with active video-games to increase physical activity and improve body composition
  Arms: exercise group with active video-games

SUMMARY:
Active video games are presented as an exercise option for children with little interest in traditional sports. The main objectives of this study are:

1. To evaluate the effects of an active video game program on cardiometabolic risk in overweight/obese children
2. to identify the effect of this intervention on physical fitness
3. to study possible changes in the sedentary lifestyles of children after the exercise program.

This is a randomized crossover study, with 2 intervention periods of 9 months each, and a 3-month period of washing. Ninetytwo children between 9 and 11 years old who are overweight or obese will be included and randomly assigned to one of the 2 homogeneous groups (control-intervention). Both groups will receive education in healthy lifestyles, and the intervention group will also follow a physical exercise program with active video games (3-4 days/week). The sessions will last between 30 and 45 minutes and will include different moderate-vigorous aerobic activities and muscular strength exercises. Body composition, physical fitness, levels of leptin, adiponectin and visfatin, lipid and ferric profiles, and markers of inflammation and metabolic risk such as insulin resistance, TNF-α, CRP, ALT, AST, gamma-GT and IL-6will be measured before and after the intervention. In addition, dietary habits (24h recalls), physical activity (accelerometers), blood pressure, waist and neck circumference, and pubertal development will be also assessed.

DETAILED DESCRIPTION:
Childhood obesity is one of the main problems in developed societies, and entails enormous expenditure for the National Health System. In addition, childhood obesity is strongly associated with adult obesity and with all types of cardiovascular and metabolic pathologies. Physical exercise has been shown to be the great non-pharmacological enemy of both childhood and adult obesity, however sport practice and adherence to it is not easy in the overweight/obese population. In this context, active video games are presented as an exercise option for children with little interest in traditional sports. The main objectives of this study are: (1) To evaluate the effects of an active video game program on cardiometabolic risk in overweight/obese children; (2) to identify the effect of this intervention on physical fitness and (3) to study possible changes in the sedentary lifestyles of children after the exercise program.

This is a randomized crossover study, with 2 intervention periods of 9 months each, and a 3-month period of washing. Ninetytwo children between 9 and 11 years old who are overweight or obese will be included and randomly assigned to one of the 2 homogeneous groups (control-intervention). Both groups will receive education in healthy lifestyles, and the intervention group will also follow a physical exercise program with active video games (3-4 days/week). The sessions will last between 30 and 45 minutes and will include different moderate-vigorous aerobic activities and muscular strength exercises. Body composition, physical fitness, levels of leptin, adiponectin and visfatin, lipid and ferric profiles, and markers of inflammation and metabolic risk such as insulin resistance, TNF-α, CRP, ALT, AST, gamma-GT and IL-6will be measured before and after the intervention. In addition, dietary habits (24h recalls), physical activity (accelerometers), blood pressure, waist and neck circumference, and pubertal development will be also assessed.

ELIGIBILITY:
Inclusion Criteria:

* children with obesity and overweight
* children with ages between 9-11 years old
* children in tanner stage I ó II

Exclusion Criteria:

* to take drugs that can affect the measurements
* menarche in girls
* contraindications or pathologies associated with exercise
* regular attendance at extracurricular activities of high energy expenditure
* diet

Ages: 9 Years to 11 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 92 (Actual)
Dates: Start 2018-11-05 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Change in fat mass during 6 months evaluated by Dual energy X-ray absorptiometry | Change from baseline in fat mass at 6 months
  Fat mass is measured by dual X-ray photon absorptiometry (DXA) using the software and pediatric reference values (Hologic Explorer, Hologic Corp., Software Latest Version, Waltham, MA).
Change in size during 6 months evaluated by a height rod to the nearest 0.1 cm (SECA 225, SECA, Hamburg, Germany). | Change from baseline in size at 6 months
  Height is measured with a height rod to the nearest 0.1 cm (SECA 225, SECA, Hamburg, Germany),
Change in size during 6 months evaluated by a 0.1 kg precision bascule (SECA 861, SECA, Hamburg, Germany) | Change from baseline in weight at 6 months
  Weight of the children is measured by a 0.1 kg precision bascule (SECA 861, SECA, Hamburg, Germany)
Change in waist and hip circumference during 6 months evaluated by an anthropometric tape following the ISAK protocol. | Change from baseline in waist and hip circumference at 6 months
  The waist and hip circumference are measured following the ISAK protocol and measurement technique with an anthropometric tape (Holtain).
Change in height jump during 6 months evaluated by countermovement jump test | Change from baseline in countermovement jump at 6 months
  Jump is measured by calculating flight height during countermoving jumps (CMJ) with a Kistler force platform.
Change in maximum manual pressure during 6 months evaluated by a manual dynamometry. | Change from baseline in dynamometry at 6 months
  Maximum manual pressure force measured by a manual dynamometry is performed with a Takei-Grip dynamometer (Espana-Romero, 2010) from 5 to 100 kg adjusting the grip to the optimal measure to develop the greatest strength as described for boys and girls
Change in knee extension isometric strength during 6 months evaluated by a strain gage. | Change from baseline in isometric knee extension strength at 6 months
  The isometric maximum force of quadriceps extension is evaluated by means of a strain gage anchored firmly to the wall and connected to a specific interface (MuscleLab); the force exerted by the subject for 10 seconds is measured and the maximum peak force is recorded.
Change in cardiorespiratory fitness during 6 months evaluated by a continuous progressive stress test | Change from baseline in cardiorespiratory fitness at 6 months
  To assess cardiorespiratory resistance, a continuous progressive test will be carried out until exhaustion, with electrocardiographic control and breath-by-breath gas analysis to measure VO2max by a maximum test with gas analyzer (Oxycon Pro, Jaeger / Viasys, Germany).
Change in the level of physical activity during 6 months evaluated by accelerometry. | Change from baseline in physical activity at 6 months
  Accelerometer measures diferent intensities of physical activity during 1 week before and after the training with videogames
Change in markers of inflammation and metabolic risk during 6 months evaluated by blood analysis | Change from baseline in markers of inflammation at 6 months
  to evaluated the biochemical analysis
Change in systolic blood pressure during 6 months evaluated by sphygmomanometer | Change from baseline in systolic blood preasure at 6 months
  Systolic blood pressure are measured, in duplicate, at rest with a sphygmomanometer (Omron M3).
Change in diastolic blood pressure during 6 months evaluated by sphygmomanometer. | Change from baseline in diastolic blood pressure at 6 months
  Diastolic blood pressure are measured, in duplicate, at rest with a sphygmomanometer (Omron M3).

CONTACTS AND LOCATIONS:
Locations (1):
- José Antonio Casajús Mallén, Zaragoza, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Comeras-Chueca C, Villalba-Heredia L, Lozano-Berges G, Matute-Llorente A, Marin-Puyalto J, Vicente-Rodriguez G, Casajus JA, Gonzalez-Aguero A. High muscular fitness level may positively affect bone strength and body composition in children with overweight and obesity. Arch Osteoporos. 2024 Jun 10;19(1):47. doi: 10.1007/s11657-024-01405-3. PMID 38856950
- [Derived] Comeras-Chueca C, Villalba-Heredia L, Perez-Lasierra JL, Lozano-Berges G, Matute-Llorente A, Vicente-Rodriguez G, Casajus JA, Gonzalez-Aguero A. Effect of an Active Video Game Intervention Combined With Multicomponent Exercise for Cardiorespiratory Fitness in Children With Overweight and Obesity: Randomized Controlled Trial. JMIR Serious Games. 2022 May 24;10(2):e33782. doi: 10.2196/33782. PMID 35471240